CLINICAL TRIAL: NCT07392398
Title: Effects of Virtual Reality Combined With Bobath Technique on Lower Limb Muscle Activity, Balance, and Motor Function in Patients With Spastic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Virtual Reality Combined With Bobath Therapy for Spastic Cerebral Palsy
Acronym: VR-BOBATH-CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, Guizhou Province (Other)
Responsible Party: Principal Investigator, Ning Li, Principal Investigator, Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, Guizhou Province
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THKTCMH-VR-BOBATH-CP-01
Record Dates: First submitted 2026-01-25; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Spastic Cerebral Palsy (sCP)
Keywords: Virtual Reality Rehabilitation; Bobath Technique; Pediatric Rehabilitation; Lower Limb Function; Balance Training; Surface Electromyography; Gross Motor Function Measure; Randomized Controlled Trial
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either a virtual reality combined with Bobath therapy group or a conventional Bobath therapy group, and outcomes will be compared between groups after a 6-week intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Combined With Bobath Therapy (Experimental): Participants in this arm will receive immersive, task-oriented virtual reality training combined with Bobath neurodevelopmental therapy. The intervention will be delivered by experienced physical therapists for 40 minutes per session, five sessions per week, over a 6-week period.
  Interventions: Behavioral: Virtual Reality Combined With Bobath Therapy
- Conventional Bobath Therapy (Active Comparator): Participants in this arm will receive conventional Bobath-based neurodevelopmental therapy without virtual reality components. The intervention frequency and duration will be the same as the experimental group, with 40-minute sessions conducted five times per week for 6 weeks.
  Interventions: Behavioral: Conventional Bobath Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Combined With Bobath Therapy — Immersive, task-oriented virtual reality training integrated with Bobath neurodevelopmental therapy, delivered by trained physical therapists. Each session will last 40 minutes and will be conducted five times per week for a total duration of 6 weeks.
  Arms: Virtual Reality Combined With Bobath Therapy
Behavioral: Conventional Bobath Therapy — Standard Bobath-based neurodevelopmental therapy provided by experienced physical therapists, without the use of virtual reality. Sessions will last 40 minutes and will be conducted five times per week for a total duration of 6 weeks.
  Arms: Conventional Bobath Therapy

SUMMARY:
Spastic cerebral palsy is a common neurodevelopmental disorder characterized by increased muscle tone, impaired balance, and limitations in motor function, particularly in the lower limbs. Conventional rehabilitation approaches such as the Bobath technique are widely used to improve posture control and movement patterns; however, patient engagement and task variability may be limited.

This randomized controlled trial aims to evaluate the effectiveness of virtual reality (VR) combined with Bobath therapy on lower limb muscle activity, balance, and gross motor function in patients with spastic cerebral palsy. Eligible participants will be randomly assigned to either a VR plus Bobath intervention group or a conventional Bobath therapy group.

The intervention will be delivered over a 6-week period, with sessions conducted five times per week. Outcome measures, including surface electromyography (sEMG), center of pressure (COP) parameters, and the Gross Motor Function Measure-88 (GMFM-88), will be assessed before and after the intervention. This study seeks to provide evidence on whether integrating VR into conventional rehabilitation can improve functional outcomes in children with spastic cerebral palsy.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized controlled trial designed to investigate the effects of virtual reality (VR) combined with Bobath therapy on lower limb muscle activity, balance, and motor function in patients with spastic cerebral palsy.

Participants aged 2 to 14 years who are diagnosed with spastic diplegic or hemiplegic cerebral palsy and classified as Gross Motor Function Classification System (GMFCS) levels I to III will be recruited. Eligible participants will be randomly allocated in a 1:1 ratio to either the experimental group or the control group.

The experimental group will receive immersive, task-oriented VR training combined with Bobath neurodevelopmental therapy. The control group will receive conventional Bobath-based rehabilitation without VR components. Both groups will undergo training sessions lasting 40 minutes per session, five sessions per week, for a total duration of 6 weeks. All interventions will be delivered by experienced physical therapists.

Primary outcomes include lower limb muscle activity assessed by surface electromyography (sEMG) of the rectus femoris, biceps femoris, tibialis anterior, and soleus muscles; balance performance evaluated using center of pressure (COP) parameters; and gross motor function measured by the Gross Motor Function Measure-88 (GMFM-88), specifically dimensions D (standing) and E (walking, running, and jumping). Assessments will be conducted at baseline and immediately after completion of the intervention period.

Secondary outcomes may include measures of participation and quality of life. Data will be analyzed using appropriate statistical methods, including repeated measures analysis of variance and covariance analysis, with a significance level set at p < 0.05.

This study aims to provide clinical evidence regarding the potential benefits of integrating virtual reality into conventional Bobath therapy for lower limb rehabilitation in children with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 14 years at the time of enrollment.
* Diagnosed with spastic cerebral palsy (spastic diplegia or spastic hemiplegia) by a qualified clinician.
* Classified as Gross Motor Function Classification System (GMFCS) levels I to III.
* Presence of lower limb spasticity with a Modified Ashworth Scale (MAS) score of at least 1.
* Ability to understand and follow simple instructions appropriate for age and cognitive level.
* Written informed consent obtained from a parent or legal guardian.

Exclusion Criteria:

* Presence of severe cognitive impairment that prevents participation in the intervention or assessments.
* Uncontrolled epilepsy or a history of frequent seizures that may interfere with the intervention.
* Severe visual, vestibular, or auditory impairments that limit safe participation in virtual reality training.
* Orthopedic surgery or botulinum toxin injection involving the lower limbs within the previous 6 months.
* Participation in other interventional clinical studies during the study period.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Lower Limb Muscle Activity Assessed by Surface Electromyography | Baseline and immediately after 6 weeks of intervention
  Lower limb muscle activity will be assessed using surface electromyography (sEMG). The sEMG amplitude and activation patterns of the rectus femoris, biceps femoris, tibialis anterior, and soleus muscles will be recorded during standardized functional tasks.
Balance Function Assessed by Center of Pressure Parameters | Baseline and immediately after 6 weeks of intervention
  Balance function will be evaluated using center of pressure (COP) measurements obtained from plantar pressure analysis. Static and dynamic balance parameters will be analyzed to assess postural control.
Gross Motor Function Measured by the Gross Motor Function Measure-88 | Baseline and immediately after 6 weeks of intervention
  Gross motor function will be assessed using the Gross Motor Function Measure-88 (GMFM-88). Dimension D (standing) and Dimension E (walking, running, and jumping) scores will be used for analysis.

SECONDARY OUTCOMES:
Overall Quality of Life Score Assessed by PedsQL Total Score | Baseline and immediately after 6 weeks of intervention
  Quality of life will be assessed using the total score of the Pediatric Quality of Life Inventory (PedsQL).
Domain-Specific Quality of Life Scores Assessed by PedsQL | Baseline and immediately after 6 weeks of intervention
  Domain-specific scores of the Pediatric Quality of Life Inventory (PedsQL), including physical, emotional, social, and school functioning, will be analyzed separately.
Attendance Rate of Scheduled Rehabilitation Sessions | Throughout the 6-week intervention period
  Attendance rate will be calculated as the proportion of attended sessions out of the total scheduled rehabilitation sessions during the intervention period.
Completion Rate of the Rehabilitation Program | Throughout the 6-week intervention period
  Completion rate will be defined as the proportion of participants who complete the full 6-week rehabilitation program as scheduled.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Principal Investigator — Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, Guizhou Province
Locations (1):
- Hongxinkang New Traditional Chinese Medicine Hospital, Tongren, Tongren, Guizhou, China

IPD SHARING:
Plan to Share IPD: Undecided